CLINICAL TRIAL: NCT02415283
Title: Evaluation of the Capability of the ¹³C-Octanoate Breath Test (OBT) Measurement to Differentiate Between Presence and Absence of HCC Determined by MRI in Patients With Chronic Liver Disease
Brief Title: OBT Measurement to Differentiate Between Presence and Absence of HCC Determined by MRI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Principal Investigator, Yongping Yang, Director of Department, Beijing 302 Hospital
Other Study IDs: HCC-MPBA-0514
Record Dates: First submitted 2015-04-09; First posted 2015-04-14 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: HCC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- HCC positive: ¹³C-Octanoate Breath Test in 50 MRI proven HCC positive patients
  Interventions: Device: ¹³C-Octanoate Breath Test
- HCC negative: ¹³C-Octanoate Breath Test in 50 MRI proven HCC negative patients
  Interventions: Device: ¹³C-Octanoate Breath Test

INTERVENTIONS:
Device: ¹³C-Octanoate Breath Test — Breath testing utilizing 13C is a safe, non-invasive means for measuring a certain pathway's metabolic rate. 13C is a stable, non-radioactive isotope which can be incorporated into a specific location within a test substrate so it would be released when the compound is metabolized by the liver. Hepatic metabolism of the compound is assessed by measuring the ratio of 13CO2/12CO2 in exhaled breath.

SUMMARY:
The Exalenz clinical investigation is a multicenter, non-randomized, study of the ¹³C-Octanoate Breath Test (OBT). The present study is a feasibility trial, which aims to evaluate the capability of the OBT to differentiate between presence and absence of HCC determined by Magnetic Resonance Imaging (MRI) in patients with chronic liver disease.

DETAILED DESCRIPTION:
1. Informed consent will be obtained from all patients prior to enrollment.
2. The trial will be conducted in compliance with this protocol, with GCP standards, and the applicable regulatory requirements.
3. This study will be cross-sectional, where patients will be enrolled on a walk in basis. Once one arm is completed the other one will be enriched in order to obtain at least 50 positive and at least 50 negative HCC subjects as defined by MRI.
4. All patients will undergo AFP and US if they do not have results within the past three months.
5. If the patient undergoes liver FNA, the biopsy results will be evaluated for the presence of HCC.
6. For all patients, a case report form will be completed.
7. All patients will undergo a physical examination, and their medical history/concomitant medications, weight, height and age will be recorded. Furthermore, recent (past 3 months) blood test results, if available, may be recorded.
8. If relevant (woman of child bearing age), a pregnancy test will be performed to rule out pregnancy when performing the breath test.
9. All MRI negative patients with low OBT results will undergo additional MRI within 6 to 12 months post OBT to rule out HCC occurrence.
10. If available, all additional MRI/CT/US results will be recorded within the patient's CRF.

ELIGIBILITY:
Inclusion Criteria:

1. Any patients with chronic liver disease at risk for HCC.
2. Age ≥ 18 years.
3. Patient has an MRI result (positive or negative for HCC) up to 3 months prior to recruitment or will be scheduled for an MRI during the trial period.
4. Patient is naïve to HCC treatment (RFA or TACE or Oral HCC treatments) since last MRI.

Exclusion Criteria:

1. Any patients with chronic liver disease at risk for HCC.
2. Age ≥ 18 years.
3. Patient has an MRI result (positive or negative for HCC) up to 3 months prior to recruitment or will be scheduled for an MRI during the trial period.
4. Patient is naïve to HCC treatment (RFA or TACE or Oral HCC treatments) since last MRI.
5. Patients currently receiving total parenteral nutrition if they have contraindications to oral drugs.
6. Women who are pregnant or breast feeding.
7. Patient taking drugs that can interfere with octanoate metabolism or can also cause NAFLD independent of the metabolic syndrome, including: corticosteroids, amiodarone, tetracycline, valproic acid, methotrexate, stavudine, zidovudine.
8. Patient, based on the opinion of the investigator, should not be enrolled into this study.
9. Patient unable or unwilling to sign informed consent.
10. Patients that are participating in other clinical trials evaluating experimental treatments or procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The proposed study will include subjects with chronic liver disease of any cause at risk for HCC with MRI results within 3 months prior to OBT or scheduled for MRI within the time frame of the study, and who meet the inclusion criteria and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-03 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
13CO2/12CO2 ratio | 60min

CONTACTS AND LOCATIONS:
Overall Officials: yongping yang, Prof, Principal Investigator — Cooperation